CLINICAL TRIAL: NCT02806206
Title: The Effect of Prucalopride on Small Bowel Transit Time in Patients Undergoing Capsule Endoscopy: A Randomized Controlled Trial
Brief Title: Prucalopride Prior to Small Bowel Capsule Endoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H16-01345
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Gastrointestinal Hemorrhage; Crohn Disease; Celiac Disease; Intestinal Diseases; Inflammatory Bowel Diseases
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Crohn Disease; Celiac Disease; Intestinal Diseases; Inflammatory Bowel Diseases | interventions — prucalopride; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Prucalopride (Experimental): A single 2 mg dose of prucalopride before ingesting the capsule endoscopy pill.
  Interventions: Drug: Prucalopride
- Drug: Placebo (Placebo Comparator): A placebo pill just before ingesting the capsule endoscopy pill.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — A single 2 mg oral dose of prucalopride will be given to each study participant just before the ingestion of the capsule endoscopy pill.
  Other Names: Restoran
  Arms: Drug: Prucalopride
Drug: Placebo — A single dose of a placebo pill will be given to each study participant just before the ingestion of the capsule endoscopy pill.
  Other Names: Sugar pill
  Arms: Drug: Placebo

SUMMARY:
Small bowel capsule endoscopy is a test used to investigate for any abnormalities in the small bowel. The small bowel is about 4 meters long. The battery time of the capsule is about 8 hours. During this time the capsule takes pictures as it passes through the small bowel. In about 15-20% of capsule tests the battery expires before the capsule passes through the entire small bowel into the colon. Incomplete tests indicate that a variable portion of small bowel was not visualized. Incomplete tests are associated with potential missing of abnormalities in the portion of small bowel that was not reached. The capsule test may often required to be repeated but the problem of incomplete examination may persist. At present no medication has been approved to increase the rate of complete capsule tests.

Prucalopride is a medication that has been approved in Canada and Europe for the treatment of chronic idiopathic constipation. Animal and human studies suggested that prucalopride may enhance the movement of the stomach and the small bowel. A recent presentation at a medical meeting suggested that prucalopride may accelerate the passage of the capsule camera through the small bowel without increasing the chance to miss a lesion in the small bowel.

The purpose of this study is to asses if the administration of a single dose of prucalopride is going to decrease the time required by the capsule to move through the small bowel.

DETAILED DESCRIPTION:
Capsule Endoscopy is now the first test to investigate for small bowel disease. Clinical conditions in which capsule endoscopy can be useful include gastrointestinal bleeding of unclear source, Crohn's disease, celiac disease and suspected small bowel tumors. Optimal diagnostic yield of the capsule endoscopy depends not only on adequate small bowel visualization, but also on the completion of small bowel examination. In approximately 15-20% of capsule studies, the capsule fails to pass through the small bowel into the colon because of the limited battery time which is about 8 hours. This means that a lesion or an abnormality can be missed in the portion of the small bowel that was not reached by the capsule. As a result, the capsule endoscopy test may often need to be repeated.

Multiple factors have been associated with the prolongation of the time required for the capsule to pass through the small bowel including hospitalization, prior small bowel surgery, diabetes and advanced age in addition to the prolongation of the time required for the capsule to pass through the stomach. Interventions to shorten small bowel transit time are required to increase capsule small bowel completion rates. At present there is no drug approved to shorten the small bowel transit time.

Prucalopride is a drug that has been approved for use in patients with chronic constipation. Prucalopride works on special receptors in the gut and stimulate the gut movement. There are basic and clinical studies suggesting that prucalopride may accelerate the movement of the stomach and the small bowel. Therefore, prucalopride may accelerate the passage of the capsule through the small bowel and increase the capsule completion rates. The investigators of this trial recently presented their experience of prucalopride use prior to capsule endoscopy at a medical meeting. Compared to a retrospective control group who did not receive prucalopride, prucalopride accelerated the passage of the capsule through the small bowel. There was no decrease in the diagnostic yield in the group who received prucalopride.

In this clinical trial, the investigators aim to investigate the effect of prucalopride on the small bowel transit time, by performing a randomized placebo controlled trial. Patients undergoing small bowel capsule endoscopy tests will be randomized to a single dose of prucalopride ingested at the time of capsule endoscopy ingestion, or a placebo pill. The primary objective of this study is to examine if the administration of a single dose of prucalopride shortens small bowel transit time compared to placebo. The secondary objectives include examining the effect of prucalopride on gastric transit time, small bowel capsule endoscopy completion rate and the capsule diagnostic yield. The placebo group is used in this clinical trial because there is no drug proven to be effective to shorten the small bowel transit time.

Based on the experience of the investigators, the average small bowel transit time for patients who were given prucalopride was 143 minutes. In the retrospective control group, the small bowel transit time was 229 minutes with a standard deviation of 90 minutes. Based on a presumed 20% minimal clinically important difference in small bowel transit time, the investigators determined a total of 122 participants will be required, equally divided between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate indication for small bowel capsule endoscopy.
* Age 19 or older.

Exclusion Criteria:

* Previous partial or complete gastric resection.
* Previous small bowel surgery in which a small bowel resection has been performed or the normal anatomy has been altered.
* Presence of ileostomy.
* The requirement for endoscopic placement of the capsule endoscopy pill because of dysphagia or gastroparesis.
* Severe renal impairment, defined by the requirement for dialysis.
* Pregnancy or breast feeding.
* Clinical or radiological suspicion of small bowel obstruction.
* Simultaneous use of a prokinetic agent within 5 days of the capsule endoscopy examination.
* Clinical hypo- or hyperthyroidism.
* Known hypersensitivity to the study drug.
* Unwillingness to sign informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Small bowel transit time | 10 hours post dose
  The calculated time from the first duodenal image to the first cecal image. The capsule images will be collected when the capsule is finished recording, approximately 10 hours post-dose.

SECONDARY OUTCOMES:
Gastric transit time | 10 hours post dose
  The calculated time from the first gastric image to the first duodenal image. The capsule images will be collected when the capsule is finished recording, approximately 10 hours post-dose.
Small bowel completion rate | 10 hours post dose
  The proportion of capsule studies in which the capsule reached the cecum. The capsule images will be collected when the capsule is finished recording, approximately 10 hours post-dose.
Diagnostic yield | 10 hours post dose
  The findings were considered diagnostic if the observed finding could explain the signs/symptoms of the patient and helped plan further management or were later confirmed by other modalities. The capsule images will be collected when the capsule is finished recording, approximately 10 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Fergal Donnellan, MD, Principal Investigator — Division of Gastroenterology, University of British Columbia; Majid Alsahafi, MD, Study Director — Division of Gastroenterology, University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No